CLINICAL TRIAL: NCT02340793
Title: Body Composition and Energy Expenditure With Total Diet Replacement During Weight Loss and Maintenance
Brief Title: BEYOND Weight Loss Study
Acronym: BEYOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN14RA448
Record Dates: First submitted 2014-12-19; First posted 2015-01-19 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Obesity
Keywords: Weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Counterweight Plus Dietary Intervention (Experimental): Weight management programme including total diet replacement with soups and shakes; approximately 800 calories/day
  Interventions: Dietary Supplement: Counterweight Plus

INTERVENTIONS:
Dietary Supplement: Counterweight Plus — A non-surgical, nutritionally replete weight management programme comprising a Total Diet Replacement Plan (TDR) of 800+ calories/day to produce a weight loss of >15kg over 12-20 weeks; followed by a structured Food Reintroduction phase for 6-8 weeks and a Weight Loss Maintenance phase; total intervention period 2 years.

SUMMARY:
National guidelines recommend 15-20% weight loss for severe and complicated obesity. Weight loss maintenance can be achieved in around 33% of patients at 12 months.

The BEYOND study will administer Counterweight Plus; a nutritionally replete Total Diet Replacement Plan (TDR) of 800+ Calories followed by structured Food Reintroduction, and Weight Loss Maintenance programmes.

The study will incorporate three work packages with the aim of:

1. examining changes in body composition with substantial (target >15kg) non-surgical weight loss (work package 1, WP1)
2. characterizing the metabolic adaptations during weight loss and maintenance (work package 2, WP2)
3. examining Rescue Packages as a method of weight re-gain prevention (work package 3, WP3).

DETAILED DESCRIPTION:
All participants will receive the Counterweight Plus dietary intervention. This consists of:

* 12-20 weeks 800+ calories/day Total Diet Replacement Plan, followed by
* 6-8 weeks Food Reintroduction, followed by
* up to 104 weeks Weight Loss Maintenance, based on maintaining daily calorie restriction.

All participants will undergo the following investigations at baseline and at regular intervals throughout the study period:

* height (baseline only)
* whole body MRI scans: total-body skeletal muscle volume and fat mass will be measured using whole-body multi-slice MRI (baseline and 12 weeks only)
* functional assessment: completion of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) (baseline and 12 weeks only)
* gait and muscle strength assessment: biomechanical gait analysis will be carried out using an 8 camera VICON system during flat walking to determine maximum flexion and extension moments for both limbs and maximum adduction and abduction moments. Muscle strength will also be directly measured of both the upper (grip strength) and lower (quadriceps and hamstrings) limb using a dynamometer and myometer (baseline and 12 weeks only)
* anthropometric measurement: body weight; waist, hip, thigh, arm and calf circumferences
* indirect calorimetry: resting metabolic rate will be measured by a computerised open-circuit ventilated hood system
* fasting blood sampling: for measurement of HbA1C, lipid profile, leptin, thyroid hormones
* gut microbiota analysis from faecal samples
* Binge Eating Disorder and Quality of Life (EQ-5D) questionnaires

Participants will receive regular support/advice from a research dietician/ nutritionist during the two year study period.

ELIGIBILITY:
Inclusion Criteria:

* confirmation from general practitioner (GP) of suitability for intervention
* written informed consent
* female
* BMI ≥30 kg/m2 and < 45kg/m2, weight<200 kg and <60 cm bore size

Exclusion Criteria:

* known illness such as heart disease, cancer, or any disability that would affect weight loss (diabetes not an exclusion) or prevent completion of the intervention
* implanted electronic devices that are MRI incompatible or MRI unsafe, ferromagnetic foreign bodies
* substance abuse
* myocardial infarction within previous 6 months
* learning difficulties and subjects having difficulty in understanding verbal or written English
* pregnant/ considering pregnancy
* patients who have required hospitalisation for depression or are on antipsychotic drugs
* people currently participating in another clinical research trial
* recent weight loss >5kg within the last 6 months
* current treatment with anti-obesity drugs
* diagnosed eating disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
WP1: change in body composition with substantial, non-surgical, weight loss | 20 weeks
  Measurement of muscle mass before and after a weight loss programme using MRI
WP1: change in body composition with substantial, non-surgical, weight loss | 20 weeks
  Measurement of fat mass before and after a weight loss programme using MRI
WP2: metabolic adaptation during weight loss and maintenance | 2 years
  Change in resting metabolic rate before and after weight loss
WP3: weight regain prevention | 2 years
  % achieving >15kg weight loss at 12 and 24 months

SECONDARY OUTCOMES:
Muscle/fat mass of specific muscle groups | 20 weeks
  Relationship between predicted muscle and fat mass with the strength of specific muscle groups (by muscle strength, gait analysis and WOMAC questionnaire)
Adherence and acceptability of Rescue Packages to Patients | 2 years
  Number of participants requiring and completing rescue packages
Metabolic adaptive effect of weight loss | 2 years
  Comparison of leptin, ghrelin and thyroid hormone levels at baseline to those during weight loss and maintenance to establish
Weight regain prevention | 2 years
  changes in BED Questionnaire Rating Score
Weight regain prevention | 2 years
  % undertaking Rescue Package during Weight Loss Maintenance
Weight regain prevention | 2 years
  rate of weight regain during Weight Loss Maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Michael EJ Lean, MA MB BChir MD, Principal Investigator — University of Glasgow
Locations (1):
- Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom